CLINICAL TRIAL: NCT07027904
Title: Immediate Implant Placement Using Xenograft as Space Filling Material Mixed With Platelet-Rich Fibrin (PRF) Versus Hyaluronic Acid in Posterior Mandible Region
Brief Title: Immediate Implant in Posterior Mandible Region
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: WASIM MHD JEHAD HALABI (Other)
Responsible Party: Sponsor-Investigator, WASIM MHD JEHAD HALABI, Bachelor's Degree of Oral and Dental Medicine, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: xenograft with (PRF)
Record Dates: First submitted 2025-05-19; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Immediate Implant With Bone Graft
MeSH Terms: interventions — Mutagenesis, Insertional

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- using xenograft as space filling material mixed with hyaluronic acid (Active Comparator): the jumping space will packed using Xenograft (cur oss , Astro star) with particle size ranging from 0.25 to 1 mm and it will be mixed with hyaluronic acid
  Interventions: Device: Implant
- xenograft (cur oss , Astro star ) mixed with Platelet-Rich Fibrin (PRF) (Experimental): the jumping space will packed using Xenograft (cur oss , Astro star) with particle size ranging from 0.25 to 1 mm and it will be mixed with Platelet-rich fibrin (PRF)
  Interventions: Device: Implant

INTERVENTIONS:
Device: Implant — The immediate implant was placed, and the surrounding cavity was filled with xenograft bone material, along with the application of hyaluronic acid or platelet-rich fibrin (PRF) to enhance healing and bone integration.

SUMMARY:
This study aims to evaluate implant stability and Width bone after placement of immediate implant and Xenograft mixed with Hyaluronic acid or with Platelet-Rich Fibrin (PRF) at posterior mandible region

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥ 18 years.

  * Both sexes.
  * Cooperative and likely to maintain good dental health.
  * Recent extraction multi roots.
  * There is a bone between (2 or 3) mm at lest from the apex of the root.

Exclusion Criteria:

* • Patients who had undergone previous extraction of all badly decayed teeth .

  * Implant placement in both healed bone and at the extraction sites in the same procedure.
  * Presence of any local or systemic factors that might contraindicate oral surgery.
  * Poor oral hygiene.
  * Conditions that complicate wound healing such as uncontrolled diabetes, smoking (10 cigarettes a day), pregnancy, a history of drug or alcohol abuse, and an inability or unwillingness to return for follow-ups after occlusal loading.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-12 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Implant secondary stability | 6 months
  Method of Measurement (Using the Osstell® Device.) -Unit of Measurement (ISQ)

SECONDARY OUTCOMES:
width bone | immediate postoperative and at 6 months
  Method of Measurement (Conebeam computed tomography (CBCT) ) -Unit of Measurement (Hounsfield unit)

IPD SHARING:
Plan to Share IPD: No